CLINICAL TRIAL: NCT03087942
Title: An Open-label, Single-dose, Parallel Group Study to Assess the Pharmacokinetics of Fevipiprant (QAW039) in Patients With End-stage Renal Disease on Hemodialysis and Optionally in Patients With Severe to Moderate and Mild Renal Impairment Compared to Matched Healthy Volunteers Including a Cross-over Assessment in End-stage Renal Disease Patients on the Effect of Dialysis on Fevipiprant Pharmacokinetics
Brief Title: Pharmacokinetics and Safety of Fevipiprant in Patients With Renal Impairment Compared to Matched Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQAW039A2107; 2016-004218-81 (EudraCT Number)
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-06

CONDITIONS: Renal Insufficiency
Keywords: end stage renal disase ESRD; dialysis effect on pharmacokinetics PK; renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — fevipiprant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): ESRD patients
  Interventions: Drug: QAW039
- Group 2 (Experimental): healthy volunteers
  Interventions: Drug: QAW39A
- Group 3 (Experimental): severe and moderate renal impaired patients
  Interventions: Drug: QAW39A2107
- Group 4 (Experimental): mild renal impaired patients
  Interventions: Drug: QAW39A2107

INTERVENTIONS:
Drug: QAW039 — 450 mg
  Other Names: fevipiprant
  Arms: Group 1
Drug: QAW39A — 450 mg
  Other Names: fevipiprant
  Arms: Group 2
Drug: QAW39A2107 — 450 mg
  Other Names: fevipiprant
  Arms: Group 3
Drug: QAW39A2107 — 450 mg
  Other Names: fevipiprant
  Arms: Group 4

SUMMARY:
The aim of the study is to assess whether renal impairment could affect fevipiprant pharmacokinetics (PK) to the extent that dosage adjustment is appropriate for this patient population.

The study also aims to determine the effect of dialysis on the fevipiprant pharmacokinetic profile as the procedure might remove a significant fraction of the drug.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the pharmacokinetic profile of fevipiprant is different in patients with renal impariment compared to healthy matched volunteers to an extent that would require an adjustment of the dosage. Data from this study will be used to guide enrollment criteria in future clinical trials and to support regulatory submission and labeling information

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects must satisfy the criteria for normal renal function as evidenced by normal Glomerular Filtration Rate (GFR): eGFR ≥ 90 mL/min/1.73m2; each healthy subject must match in age (+/- 10years), gender, smoking status, and weight (+/- 15%), a patient from the renail impaired patient groups:
* A body mass index (BMI) within the range of 18 - 36 kg/m2
* ESRD patients on hemodialysis: an glomerulo filtration rat GFR of < 15 mL/min/1.73 m2
* patients with severe renal impairment: GFR of< 30 mL/min/1.73m2 (without need of hemodialysis);
* patients with moderate renal impairment: 30 mL/min/1.73m2 ≤ eGFR < 60 mL/min/1.73m2;
* patients with mild impairment: 60 mL/min/1.73m2 ≤ eGFR < 90 mL/min/1.73m2

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* History or evidence of any inherited bilirubin disease or disorder
* subjects participating in another study
* malignancies in the past
* Hemoglobin levels below 10 g/dL at screening
* HIV positiv
* Heavy smokers (≥20 cigarettes per day)
* Liver disease, as indicated by ALT, γ-GT, AST and alkaline phosphatase which should not exceed twice the upper limit of normal and should be stable (e.g. increased liver values known from previous patient records). Serum bilirubin > 27 μmol/L (1.6 mg/dL)
* Clinically significant ECG changes and/or arrhythmias
* Chronic infection with Hepatitis B (HBV) or Hepatitis C (HCV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Plasma concentration of fevipiprant by AUClast | 68 hours post dose
  AUClast is the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
Pharmacokinetics: Plasma concentration of fevipiprant by AUCinf | 68 hours post dose
  AUCinf is the area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics: Plasma concentration of fevipiprant by Cmax | 68 hours post dose
  Cmax is the observed maximum plasma concentration following drug administration
Pharmacokinetics: Plasma contentration of fevipiprant by AUC0-68h | 68 hours post dose
  AUC0-68h is the area under the plasma concentration from time zero to time 68 hours of the last measured concentration above the limit of quantification after dosing

SECONDARY OUTCOMES:
Relationship between plasma pharmacokinetics of fevipiprant by AUClast and between eGFR as well as creatinine clearance | 68 hours post dose
  AUClast (the area under the plasma concentration time curve from time zero to the time of the last quantifiable concentration ) related to eGFR estimated by the Modification of Diet in Renal Disease (MDRD) formula, and Cockcroft-Gault (C-G) estimated creatinine clearance
Relationship between plasma pharmacokinetics of fevipiprant by AUCinf and between eGFR as well as creatinine clearance | 68 hours post dose
  AUCinf (the area under the plasma concentration time curve from time zero to infinity) related to eGFR estimated by the Modification of Diet in Renal Disease (MDRD) formula, and Cockcroft-Gault (C-G) estimated creatinine clearance
Relationship between plasma pharmacokinetics of fevipiprant by Cmax and between eGFR as well as creatinine clearance | 68 hours post dose
  Cmax (observed maximum plasma concentration following drug administration) related to eGFR estimated by the Modification of Diet in Renal Disease (MDRD) formula, and Cockcroft-Gault (C-G) estimated creatinine clearance
Pharmacokinetics of the metabolite CCN362 by AUClast | 68 hours post dose
  AUClast is the area under the plasma concentration time curve from time zero to the time of the last quantifiable concentration
Pharmacokinetics of the metabolite CCN362 by AUCinf | 68 hours post dose
  AUCinf is the area under the plasma concentration time curve from time zero to infinity
Pharmacokinetics of the metabolite CCN362 by Cmax | 68 hours post dose
  Cmax is the observed maximum plasma concentration following drug administration
Pharmacokinetics: plasma concentration of fevipiprant in patients with End Stage Renal Disease (ESRD) | 68 hours post dose
  Partial AUCs (AUCt1-t2) covering the time interval of dialysis, Cmax and total AUCs (AUC0-68h and/or AUCinf) will be compared
urinary excretion of fevipiprant and metabolite in patients with renal impairment compared to healthy controls | 24 hours post dose
  Renal clearance (CLr) and fraction of dose excreted in urine for fevipiprant and metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Orlando, Florida, United States
- Novartis Investigative Site, Grünstadt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CQAW039A2107 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17506
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=289